CLINICAL TRIAL: NCT02119117
Title: Blastocyst Aneuploidy Rates From Advanced Maternal Age Patients Supplemented With Coenzyme Q10 (CoQ10) Versus Those That Are Not: a Pilot Study
Brief Title: Aneuploidy Rates in Advanced Maternal Age Patients Supplemented With Coenzyme Q10 (CoQ10) Versus Those That Are Not: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive Endocrinology Associates of Charlotte (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: REACh-002
Record Dates: First submitted 2014-04-14; First posted 2014-04-21 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Mitochondrial DNA; Aneuploidy
Keywords: mtDNA; aneuploidy; IVF; blastocyst; COQ10
MeSH Terms: conditions — Aneuploidy | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sugar pill (Placebo Comparator): Group 2 will receive a placebo of CoQ10
  Interventions: Dietary Supplement: Placebo
- CoQ10 (Experimental): Patients will be divided into 2 groups. Group 1 will be treated with an oral supplement, 125 mg/twice daily of CoQ10 (NeoQ10, Theralogix, Rockville, Maryland, USA) for 3 months prior to IVF. This dosage will equate to a Cmax of 6.89 ug/ml (Liu and Artmann, 2009).
  Interventions: Dietary Supplement: CoQ10

INTERVENTIONS:
Dietary Supplement: CoQ10 — This is a dietary supplement which will be administered daily to the patient for 3 months prior to IVF
  Arms: CoQ10
Dietary Supplement: Placebo — This is a placebo which will be administered daily to the patient for 3 months prior to IVF.
  Arms: sugar pill

SUMMARY:
Pregnancy rates for women over 35 years old are significantly lower when compared to younger women. One of the causes for this decrease is believed to be chromosomal aneuploidy. Chromosomal aneuploidy is a natural phenomena and occurs in women of every age and has been implicated in spontaneous miscarriages, and preimplantation embryo wastage (Hassold and Hunt, 2001).

As maternal age increases, so too does the incidence of chromosomal aneuploidy. Embryo quality from older patients undergoing IVF tends to be reduced and associated with higher rates of chromosomal abnormalities when compared to good quality embryos (Munne et al., 1995).

Chromosomal aneuploidy derives from the improper segregation of chromosomes during preimplantation development. The process of segregation, or mitosis, includes synthesis of the complete genome, equal division of chromosomes to opposite poles by the spindle apparatus, and separation of the two cells by cytokinesis, yielding two chromosomally identical cells. The entire process of cellular and genetic replication requires energy in the form of adenosine tri phosphate (ATP). ATP is mainly produced in mitochondria in the process known as the electron transport chain (ETC). There are many important molecules required for ATP production, CoQ10 can act as the appropriate carrier of electrons through the ETC. When a deficiency in CoQ10 is present, ATP production is decreased resulting in aneuploidy (Bentov et al., 2013). Similarly, research has shown that chromosome alignment and spindle formation are affected by mtDNA copy number (Ge et al., 2012). It has also been shown that the transfer of ooplasm from young, healthy oocyte donors into oocytes of women with repeated embryonic failure has result in children with subsequent mitochondrial heteroplasmy (Cohen et al., 1998).

CoQ10 concentrations have been shown to decrease as age increases (Bentov et al., 2011). Consequently, the decrease in CoQ10 concentrations seen in older women may cause an increase in chromosomal aneuploidy in subsequent embryos (Bentov et al., 2013). In this pilot study, we test the hypothesis that the supplementation of CoQ10 prior to an IVF cycle can increase mitochondrial DNA activity and possibly decrease chromosomal aneuploidy in AMA patients.

DETAILED DESCRIPTION:
Brief Summary

ELIGIBILITY:
Inclusion Criteria:

1. 36-42 years old
2. Must present with an AMH level ≤2.0 ng/mL
3. 1st cycle of IVF treatment
4. Antral follicle count >5 and <20

Exclusion Criteria:

1. BMI >39
2. Active smoker
3. Blood serum baseline level of CoQ10 ≥2.20 µg/mL
4. Prior use of CoQ10
5. Type II diabetes mellitus

Ages: 36 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Embryo mitochondrial DNA (mtDNA) | mtDNA levels will be assesed from day 5 or day 6 blastocysts

SECONDARY OUTCOMES:
preimplantation chromosomal aneuploidy | aneuploidy rates will be measured utilizing SNP array from day 5 and day 6 blastocysts

CONTACTS AND LOCATIONS:
Overall Officials: Jack L Crain, MD, Principal Investigator — Reproductive Endocrinology Associates of Charlotte
Locations (1):
- REACh, Charlotte, North Carolina, United States